CLINICAL TRIAL: NCT04585633
Title: Postoperative Risk Prediction Score After Elective Intracranial Neurosurgery Operation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation Resident Doctor, Trakya University
Other Study IDs: TÜTF-BAEK 2020/136
Record Dates: First submitted 2020-08-04; First posted 2020-10-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Brain Tumor; Post-Op Complication; Anesthesia
Keywords: craniotomy; Quality of Recovery; post-operative; risk prediction score; anesthesia recovery
MeSH Terms: conditions — Brain Neoplasms; Postoperative Complications | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Risk: no complication develop within 30 days after the operation and high GOS value
  Interventions: Other: Quality of Recovery-15; Other: Glasgow Result Scale; Other: Risk Factors
- High Risk: complication or complications develop within 30 days after the operation and low GOS value
  Complications:
  * Moderate to severe intracerebral hemorrhage confirmed in a brain CT scan (Midline shift in brain imaging ≥ 3 mm),
  * İntracranial hypertension requiring post op surgical drainage,
  * Status epilepticus or seizures,
  * The need for tracheal intubation or use of mechanical ventilation after surgery,
  * Decrease in GKS,
  * Unmanageable agitation that requires restriction or sedation,
  * Need for respiratory failure and oxygen therapy,
  * Unexpected serious motor deficit
  * Died
  Interventions: Other: Quality of Recovery-15; Other: Glasgow Result Scale; Other: Risk Factors

INTERVENTIONS:
Other: Quality of Recovery-15 — Quality of Recovery-15 is a scale consisting of 15 questions indicating the recovery quality of the patient after anesthesia and a score between 0-150.
  Other Names: QoR-15
Other: Glasgow Result Scale — Glasgow Outcome Scale; It is a scale developed to categorize people suffering from head trauma or non-traumatic acute brain injury into broad outcome categories. It shows postoperative mortality and morbidity of patients who underwent intracranial surgery.
  Other Names: GOS
Other: Risk Factors — Pre-operative: medical histories, drugs used, demographic features, additional diseases, ASA class, pre-operative routine parameters, operation history, GCS, tumor histology, location, dimensions and intracerebral radiological data, laboratory values Intraoperative; hemodynamic data of patients; highest and lowest values of heart rate, diastolic, systolic and mean arterial pressures, fluid and blood products given, anesthetic and other drugs administered, duration of anesthesia, duration of surgery, surgical position, blood loss, urine output and blood gas samples Post-operation; extubation time, MAS score, use of mechanical ventilation, post-operative complications, hemodynamic data, blood gas data

SUMMARY:
The aim of our study is to prevent unnecessary intensive care unit hospitalizations by developing a scoring system to detect low-risk patients after elective intracranial neurosurgery operation.

DETAILED DESCRIPTION:
In this study, the data of patients who are planned to undergo craniotomy by neurosurgery will be collected as a file scan (medical histories, drugs used, demographic features, additional diseases, ASA class, pre-operative routine parameters, operation history, GCS, tumor histology, location, dimensions and intracerebral radiological data, laboratory values). The pre-operative Quality of Recovery-15 (QoR-15) score will be recorded before the patient is taken into operation. Intraoperative; hemodynamic data of patients; highest and lowest values of heart rate, diastolic, systolic and mean arterial pressures, fluid and blood products given, anesthetic and other drugs administered, duration of anesthesia, duration of surgery, surgical position, blood loss, urine output and blood gas samples will be written from the anesthesia document after the operation is over. For the study, the application of the anesthesiologist for the patient will not be interfered. After the operation; extubation time, MAS score, use of mechanical ventilation, post-operative complications (moderate to severe intracerebral hemorrhage on brain CT, intracranial hypertension requiring post op surgical drainage, development of status epilepticus or seizures, the need for tracheal intubation and mechanical ventilation after surgery, decrease in GKS, unmanageable agitation that requires restriction or sedation, need for respiratory failure and oxygen therapy, serious motor deficit and exitus) will be recorded in the service where the patient is sent. The post-operative QoR-15 score will be calculated 24 hours after the operation. Pre-operative and post-operative calculated scores of the patient will be evaluated and anesthesia recovery score will be created. With this recovery score, post-operative mortality and morbidity estimates will be made. The length of hospital stay of the patient will be recorded. Glasgow Result Scale (GOS) score will be determined 30 days after the patient operation. In this way, 1 month morbidity and mortality of the patient will be evaluated. The collected results will be statistically associated with anesthesia recovery and operation complications.

As a result, in our study; post-operative risk prediction score will be created in patients undergoing intracranial surgery with elective craniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. To undergo intracranial operation with elective craniotomy
2. No history of congestive heart failure
3. No kidney and liver dysfunction
4. Not pregnant
5. To be over 18 years old

Exclusion Criteria:

1. To undergo an intracranial operation with emergency craniotomy
2. Patients with a history of congestive heart failure
3. Patients with kidney and liver dysfunction
4. Pregnant patients
5. Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include intracranial operations performed by craniotomy in a 2-year period by Trakya University Faculty of Medicine, Department of Neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 | score change before surgery and 24 hours after surgery
  Quality of Recovery-15 is a scale consisting of 15 questions indicating the recovery quality of the patient after anesthesia and a score between 0-150.

SECONDARY OUTCOMES:
Complication | during the hospital stay
  the development of complication or complications during hospitalization
  Complications:
  * Moderate to severe intracerebral hemorrhage confirmed in a brain CT scan (Midline shift in brain imaging ≥ 3 mm),
  * İntracranial hypertension requiring post op surgical drainage,
  * Status epilepticus or seizures,
  * The need for tracheal intubation or use of mechanical ventilation after surgery,
  * Decrease in GKS,
  * Unmanageable agitation that requires restriction or sedation,
  * Need for respiratory failure and oxygen therapy,
  * Unexpected serious motor deficit
  * Died
Glasgow Outcome Scale | 30th day after the operation (1 time)
  Glasgow Outcome Scale; It is a scale developed to categorize people suffering from head trauma or non-traumatic acute brain injury into broad outcome categories. It shows postoperative mortality and morbidity of patients who underwent intracranial surgery. Glasgow Outcome Scale is a five-point scale. 1 point is considered death and five points as good recovery. As the score increases, morbidity and mortality decrease.

CONTACTS AND LOCATIONS:
Overall Officials: SEVTAP HEKİMOĞLU ŞAHİN, Professor, Principal Investigator — Trakya University; ONUR KÜÇÜK, Resident, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No